CLINICAL TRIAL: NCT00453050
Title: Laser and TLR-Agonist Immunotherapy: A Novel Autologous Melanoma Vaccine Study
Brief Title: Imiquimod and Laser Therapy With or Without a Green Dye in Treating Patients With Stage III or Stage IV Melanoma That Has Spread to Other Parts of the Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000536471; OU-12576; OU-ISPI
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2008-11

CONDITIONS: Melanoma (Skin); Metastatic Cancer
Keywords: stage III melanoma; stage IV melanoma; skin metastases
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Imiquimod; Flow Cytometry; Immunologic Techniques

INTERVENTIONS:
Drug: imiquimod
Drug: indocyanine green solution
Other: flow cytometry
Other: immunologic technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Biological therapies, such as imiquimod, may stimulate the immune system in different ways and stop tumor cells from growing. Laser therapy uses light to kill tumor cells. Giving imiquimod together with laser therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects of imiquimod and laser therapy with or without a green dye in treating patients with stage III or stage IV melanoma that has spread to other parts of the skin.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity of in situ photoimmunotherapy comprising imiquimod and infrared laser therapy with or without indocyanine green in patients with stage III or IV melanoma and cutaneous metastases.
* Determine the complete systemic and local response rates in patients treated with this regimen.

Secondary

* Determine the effect of this treatment on immunologic parameters in these patients.

OUTLINE: This is a prospective, open-label, pilot study.

Patients undergo in situ photoimmunotherapy (ISPI) comprising topical imiquimod twice daily on days 1-42 and infrared laser therapy (with or without indocyanine green) on days 14 and 28. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

Blood is collected at baseline, prior to ISPI, 24 hours after ISPI, and at week 6. Samples are examined for cytokine response, CD8 T-cell activation and regulatory T-cell assays (by flow cytometry), and antibody response (by western blot).

After completion of study treatment, patients are followed monthly for 3 months and then every 3 months for up to 2 years.

PROJECTED ACCRUAL: A total of 70 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma meeting the following criteria:

  * Stage III or IV disease

    * Stage IV disease without observable, surgically unresectable metastases beyond the immediate treatment site allowed
  * Presence of 1 or more cutaneous metastases ≤ 3 cm in size

    * Diffuse areas of tumor involvement can be used to qualify for the study if these areas involve primarily the epidermis and/or dermis and are less than 3 cm in thickness
* No uncontrolled brain metastases

  * Treated brain metastases that are stable for 3 months allowed at the investigator's discretion

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 4 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after study completion
* No known allergy to any drugs used during study treatment
* No unstable medical illness
* Not immunosuppressed

  * Patients immunosuppressed due to disease (e.g., HIV positive) allowed

PRIOR CONCURRENT THERAPY:

* No systemic steroids or any other immunosuppressive medications within the past month
* No chemotherapy within the past 4 weeks
* No radiotherapy to the treatment site within the past 4 weeks

  * Palliative radiotherapy to sites other than cutaneous treatment and assessment sites allowed
* No concurrent immunosuppressive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-03; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Toxicity and tolerability by CTCAE version 3.0
Complete systemic and local response rates at 16 months

SECONDARY OUTCOMES:
Immunologic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Mark Naylor, MD, Study Chair — University of Oklahoma
Locations (1):
- Oklahoma University Cancer Institute, Tulsa, Oklahoma, United States

REFERENCES:
- [Background] Li X, Naylor MF, Le H, Nordquist RE, Teague TK, Howard CA, Murray C, Chen WR. Clinical effects of in situ photoimmunotherapy on late-stage melanoma patients: a preliminary study. Cancer Biol Ther. 2010 Dec 1;10(11):1081-7. doi: 10.4161/cbt.10.11.13434. Epub 2010 Dec 1. PMID 20890121
- [Background] Naylor MF, Chen WR, Teague TK, Perry LA, Nordquist RE. In situ photoimmunotherapy: a tumour-directed treatment for melanoma. Br J Dermatol. 2006 Dec;155(6):1287-92. doi: 10.1111/j.1365-2133.2006.07514.x. PMID 17107404